CLINICAL TRIAL: NCT06636110
Title: Piloting of JUN to Enhance Self-Efficacy Pregnant Women
Brief Title: Piloting JUN_Pregnancy Mobile Medical App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The University of Texas at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000755
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Pregnancy
Keywords: Community Supervision; Criminal Justice Oversight; Jun App

STUDY DESIGN:
Intervention Model Description: 1:1 selection of pregnant women with and without criminal justice oversight. There will be further random selection of a sub-sample (n=20) (n=10 with and n=10 without criminal justice oversight to interview using Health Belief Model (HBM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pregnant without Criminal Justice Oversight (Experimental): Pregnant women who are without criminal justice oversight
  Interventions: Device: Jun mHealth app
- Pregnant with Criminal Justice Oversight (Experimental): Pregnant women who are under Community Supervision (CS), on probation or parole with criminal justice oversight
  Interventions: Device: Jun mHealth app

INTERVENTIONS:
Device: Jun mHealth app — The intervention will be a mHealth app, JUN, across 3 months during pregnancy.
  Other Names: Mobile Medical Health App

SUMMARY:
This research activity looks at the safety of an investigational intervention, a mobile health (mHealth) app called JUN, that uses artificial intelligence (AI) to track symptoms and give time-sensitive feedback to pregnant women.

JUN is an intervention being developed to provide education and assist with decision making during pregnancy.

The researchers hope to learn differences in how effectively the participant use of the app is amongst women with and without criminal justice oversight such as adult probation or parole.

DETAILED DESCRIPTION:
In this proposed pilot study, the investigators will use mixed methods to examine differences across three months among pregnant women. Sampling will be within three ethnically and geographically diverse sites, Texas, Oregon, and Minnesota to determine if there are differences in self-efficacy amongst pregnant women on Community Service (CS) compared to pregnant women without criminal justice oversight.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female 18-50 years
2. Within first 6 months of pregnancy
3. Either on community supervision or without criminal system involvement
4. Located in Texas, Minnesota or Oregon

Exclusion Criteria:

1. Individuals who do not identify as women
2. Later pregnancy, beyond the first 6 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women in their first 6 months of pregnancy
Enrollment: 50 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Self Rated Abilities for Health Practice (SRAHP) | Baseline to Post-Intervention survey (approximately 3 months)
  The Self Rated Abilities for Health Practices Scale (SRAHP) is a 28-item, 5-point scale to measure self-perceived ability to implement health-promoting behaviors. SRAHP contains four subscales: Exercise, Nutrition, Responsible Health Practice, and Psychological Well Being. Each subscale has seven items. Respondents are asked to rate the extent to which they are able to perform health practices related to these four domains. An example of an item from the Health Practices subscale is "I am able to get help from others when I need it." Items are rated from 0 (not at all) to 4 (completely). Ratings for each subscale are summed to yield subscale scores. Subscale scores are summed to obtain a total score. Total scores range from 0-112. Higher scores indicate greater self-efficacy for health practices.
JUN mHealth app Timing | Month 1 to Month 3
  Timing of use of JUN app.
JUN mHealth app Frequency | Month 1 to Month 3
  Frequency of use of the JUN app

SECONDARY OUTCOMES:
Accountable Health Communities Health-Related Social Needs Screening (AHC HRSN) | Baseline to Post-Intervention survey (approximately 3 months)
  There are five core domains of the AHC HRSN Screening Tool: (1) living situation, (2) food, (3) transportation, (4) utilities, and (5) safety. For each domain, if the participant answers yes to one of the items, it is a positive screen. There is not a total score for this measure. Rather, it assesses what participants have and do not have.
Sigma-Related Rejection Scale | Baseline to Post-Intervention survey (approximately 3 months)
  A 9 item scale which uses multiple answer formats. The Stigma-Related Rejection Scale (SRS) (or its variations, like the Substance Abuse version) is a survey measuring interpersonal stigma and rejection experiences, with higher scores indicating greater perceived stigma and rejection.
  The SRS assesses the ongoing experiences of personal rejection related to enacted stigma, focusing on how individuals with mental health conditions or substance abuse problems perceive and experience stigma in their daily lives. Items are typically scored on a scale of 1 to 7, with higher scores indicating greater agreement with the statement and thus, higher levels of perceived rejection.
Abuse Assessment Screening tool (AAS) | Baseline to Post-Intervention survey (approximately 3 months)
  This five-item tool detects abuse perpetrated against childbearing women with a sensitivity of 93%-94% and specificity of 55%-99% related to the question specific to abuse during pregnancy (e.g., "Since you were pregnant, have you been slapped, kicked, or otherwise physically hurt by someone," Within the past year, has anyone forced you to have sexual activities?"). Evidence: Women with SUD often live in potentially abusive or violent environments, which can negatively affect their perinatal health and may lead to a return to using illicit substances. Items 1 and 5 are answered yes/no; if items 2, 3, or 4 are answered yes, participant is asked to indicate category of abuser (Circle all that apply: husband, ex-husband, boyfriend, stranger, other, multiple); for items 2 and 3, participants are asked to mark the area of injury on a body map.
  For each violence incident, items are scored based on severity of (1-6)ǂ Cutoff for IPV: Affirmative response to ≥1 item(s)
Patient Health Questionnaire (PHQ) | Baseline to Post-Intervention survey (approximately 3 months)
  Patient Health Questionnaire (PHQ2) measures the frequency and severity of depressed mood, anhedonia, and anxiety in the past weeks (e.g., "Over the last two weeks, how often have you been bothered by the following problems…feeling down, depressed, or hopeless?"). Responses are summed across items to yield a total score (e.g., cut-off scores >3 are considered elevated). PHQ-2 has 2 questions scored on a scale of 0-3 with a total score of 0-6. A score of 3 or higher indicates a need for further evaluation.
Generalized Anxiety Disorder (GAD2) | Baseline to Post-Intervention survey (approximately 3 months)
  Patient Generalized Anxiety Disorder Survey (GAD2) measures the frequency and severity of depressed mood, anhedonia, and anxiety in the past weeks (e.g., "Over the last two weeks, how often have you been bothered by the following problems…feeling down, depressed, or hopeless?"). Responses are summed across items to yield a total score (e.g., cut-off scores >3 are considered elevated).
  GAD-2 has 2 questions scored on a scale of 0-3 with a total score of 0-6. A score of 3 or higher needs further diagnostic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Allison Ihle, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
No personally identifying data is anticipated to be recorded from human subjects, neither through survey responses or other interactions.
  The PI, Co-PIs, researchers, and staff plan to make all data generated from this IIMS proposal freely available to the research community after publication. Through the freedom of information act, the data in the publications and the raw data documents will be made available upon written request to the laboratory. Should intellectual property be generated which requires a patent, we will ensure that the technology (materials and data) remains widely available to research community in accordance with the NIH Principles and Guidelines referenced above.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of this project's period, appropriate plans will be made to maintain data stored on UTHSCSA servers or otherwise upload it to a publicly-available repositor.